CLINICAL TRIAL: NCT02522403
Title: Application of Laser Acupuncture in Rehabilitating Patients With Distal Radius Fracture
Brief Title: Acupuncture in Distal Radius Fracture Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Autonoma de Nuevo Leon (Other)
Responsible Party: Principal Investigator, Carlos A Acosta-Olivo, MD, PhD, Universidad Autonoma de Nuevo Leon
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: OR15-010
Record Dates: First submitted 2015-08-06; First posted 2015-08-13 (Estimated); Results first posted 2018-10-19 (Actual); Last update posted 2018-10-19 (Actual); Status verified 2017-12

CONDITIONS: Colles´ Fracture; Radius Fracture
Keywords: distal radius fracture; laser acupuncture; rehabilitation
MeSH Terms: conditions — Colles' Fracture; Radius Fractures; Wrist Fractures | interventions — Rehabilitation; Physical Therapy Modalities; Medicine, Chinese Traditional

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Rehabilitation (Active Comparator): The investigators will be apply laser acupuncture for the rehabilitation of the wrist and hand of the patients, with the laser device in an off position, plus exercise of wrist flexion, extension, cubital and radial deviation, pronation and supination of the forearm. The investigators will be use ten different acupuncture points for treat this patients.
  Interventions: Procedure: Rehabilitation
- Low Lever Laser acupuncture (Experimental): The investigators will utilize an low level laser therapy device apply into each acupuncture point. Ten acupuncture points will be used. Each acupuncture point will be irradiated for 30 seconds at 8,000 Hz.
  Interventions: Device: Low Lever Laser acupuncture

INTERVENTIONS:
Procedure: Rehabilitation — The investigators will be apply fake laser therapy in the patients with distal radius fracture, with the device in an off position; plus the patients will be teaching to do rehabilitation exercise in flexion, extension, pronation and supination of the wrist and forearm, and to do cubital and radial deviation exercise. The investigators delivered to all patients a graphic demonstration of the exercise
  Other Names: Physical therapy
  Arms: Rehabilitation
Device: Low Lever Laser acupuncture — The investigators will be used a low lever laser device, to apply in ten selected acupuncture points, each point will be irradiated for 30 seconds at 8000 Hz, this therapy is useful for tissue regeneration and stimulate the acupuncture points, plus an antinociceptive effect.
  Other Names: Chinese traditional medicine; Needles Diller & Diller
  Arms: Low Lever Laser acupuncture

SUMMARY:
The patients with distal radius fracture treated with immobilization (cast) and percutaneous pinning it will be to able to participate in this randomized trial. The investigators will be able to determine if the laser acupuncture is a good therapy for the rehabilitation in this type of patients. And if they are more comfortable to begin his rehabilitation exercise after the application of this therapy

DETAILED DESCRIPTION:
Distal radius fractures are very common, ranging between 17 and 20% of all diagnosed fractures, and are the most common fractures treated by orthopedic surgeons in adult patients. It is defined as a fracture of the distal radius, which is less than 2.5 cm from the radiocarpal joint. Usually it is the result of falling on the outstretched hand. These fractures occur in all age groups and a bimodal distribution is observed with a peak incidence predominantly young adult patients and another peak in older women.

In order to achieve successful functional results in distal radius fracture both an adequate treatment and timely and specific rehabilitation are required. The distal radius fracture guidelines generally indicate that rehabilitation therapy should begin at four to six weeks post injury or surgery after cast or external fixator is removed initiating passive/active ranges of motion exercises for the fingers, wrist and forearm. Patients are encouraged to use the wrist at home for light activities. At nine to 12 weeks post injury patients can initiate grip strengthening.

There is limited available literature on the effect of acupuncture in the treatment of fractures. Two case reports claim to have achieved an acceleration of bone healing and pain management of patients with proximal humerus fracture when treated with a combination of acupuncture, electro-acupuncture and herbal medicine. Another study concluded that electroacupuncture plus radiation therapy with infrared rays and passive exercises was clearly superior to therapy with only exercises after surgery for humerus fracture.

There is a modality of acupuncture using low level laser therapy, which is useful for tissue regeneration in general and to stimulate acupuncture points. Current clinical research has confirmed the therapeutic usefulness of laser acupuncture in and equine laminitis and in humans in treating myofascial pain, tennis elbow, knee osteoarthritis and other musculoskeletal diseases.

The low level laser therapy, is a type of noninvasively phototherapy that has been shown to modulate various biological processes depending on the power density, wavelength and frequency. A recent study using rats showed that laser stimulation of acupuncture point (located in the leg) caused a significant antinociceptive effect controlling the behavior induced in rats caused by pain after peritoneal injection of acetic acid and injection of formalin in rat paws. The effect is mediated by activation of the opioidergic and serotoninergic systems (5HT-1 and 5HT-2A receptors).

Investigators will try to determine whether laser acupuncture has a positive effect on the rehabilitation of patients with distal radius fracture and to establish a safe therapy without adverse effects that may alleviate pain and restore the functionality of the joint as soon as possible.

This study will be a prospective, longitudinal, randomized, double-blind trial which will include 32 volunteers. All patients with a diagnosis of distal radius fracture type 23-A2, A3, B1, and B2 of the Orthopedic Trauma Association classification that comply with the inclusion criteria will be included. Patients will be randomly assigned to one of two groups: control or experimental group.

The sessions will start as soon as the patient has their cast removed. Control group will receive conventional rehabilitation exercises and "fake" laser acupuncture (device turned off). Experimental group A will receive treatment with conventional rehabilitation plus real laser acupuncture on the following points: bilateral Hegu (IG4), ipsilateral Yangxi (IG5), ipsilateral Yangchi (SJ4), ipsilateral Yanggu (ID5), ipsilateral Waiguan (SJ15), ipsilateral Daling (PC7), contralateral Taixi (R3), contralateral Shenmai (V62) and contralateral Kunlun (V60). All patients will receive a total of 10 sessions with a frequency of 3 times a week. The laser that will be used in this study is a low level laser therapy device (980nm, 50 mW). Each acupuncture point will be irradiated for 30 seconds at 8,000 Hz.

All patients will undergo clinical evaluation to assess improvement using the Patient-Rated Wrist Evaluation Scale. Patients also will be evaluated with the Visual Analogue Scale. The investigators will also measure improvement in range of motion of the wrist (flexion, extension, radial deviation, ulnar deviation, pronation and supination) and grip strength.

The first assessment will be made right before starting rehabilitation and acupuncture, the day of the 5th session, again on the day of the 10th session and finally one week after completing the 10 sessions. All evaluations should be performed by blinded investigator. The investigators will compare the two groups to determine the degree of improvement with each treatment modality used.

ELIGIBILITY:
Inclusion Criteria:

* Distal radius fracture treated with percutaneous pinning and plaster
* Type A2, A3, B1 and B2 of the Orthopedic Trauma Association classification

Exclusion Criteria:

* Rheumatoid arthritis
* Ipsilateral fractures
* Psychiatric illness
* Previous wrist fracture or surgery
* Cancer

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2015-08; Primary Completion 2016-06 (Actual); Study Completion 2016-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Carlos Acosta-Olivo, MD, PhD, Principal Investigator — Universidad Autonoma de Nuevo Leon
Locations (1):
- Universidad Autonoma de Nuevo Leon, Monterrey, Nuevo León, Mexico

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Tahririan MA, Javdan M, Motififard M. Results of pronator quadratus repair in distal radius fractures to prevent tendon ruptures. Indian J Orthop. 2014 Jul;48(4):399-403. doi: 10.4103/0019-5413.136275. PMID 25143645
- [Background] Wei XM, Sun ZZ, Rui YJ, Song XJ. Minimally invasive plate osteosynthesis for distal radius fractures. Indian J Orthop. 2014 Jan;48(1):20-4. doi: 10.4103/0019-5413.125483. PMID 24600058
- [Background] Smith DW, Brou KE, Henry MH. Early active rehabilitation for operatively stabilized distal radius fractures. J Hand Ther. 2004 Jan-Mar;17(1):43-9. doi: 10.1197/j.jht.2003.10.006. PMID 14770137
- [Background] Luo KM, Hou Z, Yang L. [Observation on therapeutic effect of electroacupuncture on activity disturbance of the shoulder joint after operation of fracture]. Zhongguo Zhen Jiu. 2008 Oct;28(10):727-9. Chinese. PMID 18972728
- [Background] Erthal V, da Silva MD, Cidral-Filho FJ, Santos AR, Nohama P. ST36 laser acupuncture reduces pain-related behavior in rats: involvement of the opioidergic and serotonergic systems. Lasers Med Sci. 2013 Sep;28(5):1345-51. doi: 10.1007/s10103-012-1260-7. Epub 2013 Jan 5. PMID 23291880

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Rehabilitation | Low Lever Laser Acupuncture
Started | 17 | 19
Completed | 13 | 13
Not Completed | 4 | 6
Not completed — Lost to Follow-up | 2 | 2
Not completed — Withdrawal by Subject | 2 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Rehabilitation | Low Lever Laser Acupuncture | Total
Number analyzed (Participants) | 13 | 13 | 26
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 10 | 12 | 22
  >=65 years | 3 | 1 | 4
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.2 (14.7) | 53.2 (9.7) | 54.8 (13.07)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 8 | 17
  Male | 4 | 5 | 9
Region of Enrollment [Number; unit: participants]
  Mexico | 13 | 13 | 26
Patiet-Rated Wrist Evaluation (PRWE) [Mean (Standard Deviation); unit: units on a scale] — The PRWE assesses pain and the inability to perform daily acitivities. Is a 15-item questionnaire designed to measure wrist pain and disability in activities of daily living. It yields a score of 0 to 100, with lower scores indicanting better performance.
  units on a scale | 70.9 (13.6) | 69.1 (12.2) | 70.1 (12.7)
Visual Analog Scale (VAS) [Mean (Standard Deviation); unit: units on a scale] — The VAS has a score of 0 to 10. The lowest score (0) represents the absence of pain, while the highest score (10) corresponds to the maximum pain possible.
  units on a scale | 5.0 (2.2) | 5.9 (1.7) | 5.5 (2.0)
Wrist Mobility [Mean (Standard Deviation); unit: degrees] — The degrees of wrist mobility in flexion, extension, pronation, supination, and radial and ulnar deviation were measured in all patients.
  degrees
    Flexion | 33.3 (18.6) | 34.2 (10.5) | 33.8 (14.9)
    Extension | 14.9 (15.1) | 22.0 (14.4) | 18.5 (14.9)
    Pronation | 44.2 (23.2) | 54.8 (25.2) | 49.5 (24.4)
    Supination | 40.3 (21.2) | 42.6 (21.3) | 41.5 (20.9)
    Ulnar Deviation | 15.7 (6.8) | 20.0 (7.6) | 17.9 (7.4)
    Radial Deviation | 7.1 (5.5) | 4.6 (4.1) | 5.9 (5.0)

OUTCOME MEASURES:

1. Primary Outcome: Patient-Rated Wrist Evaluation (PRWE)
Description: The PRWE assesses pain and the inability to perform daily acitivities. Is a 15-item questionnaire designed to measure wrist pain and disability in activities of daily living. It yields a score of 0 to 100, with lower scores indicanting better performance.
  Only the final results of the study are reported.
Time Frame: 6 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Rehabilitation | Low Lever Laser Acupuncture
Number analyzed (Participants) | 13 | 13
units on a scale | 30.5 (22.5) | 15.2 (11.9)

2. Secondary Outcome: Wrist Mobility
Description: The degrees of wrist mobility in flexion, extension, pronation, supination, and radial and ulnar deviation were measured in all patients.
  Only the final measures of movements of the study are reported.
Time Frame: 6 weeks
Measure: Mean (Standard Deviation); unit: degrees
Arm/Group | Rehabilitation | Low Lever Laser Acupuncture
Number analyzed (Participants) | 13 | 13
degrees
  Flexion | 39.8 (18.1) | 60.2 (18.9)
  Extension | 41.1 (20.6) | 52.6 (13.0)
  Pronation | 80.0 (9.3) | 88.4 (3.1)
  Supination | 67.6 (22.5) | 76.1 (13.7)
  Cubital deviation | 27.0 (9.8) | 31.3 (6.8)
  Radial deviation | 10.3 (5.1) | 18.0 (5.9)

3. Secondary Outcome: Visual Analogue Scale (VAS)
Description: The VAS has a score of 0 to 10. The lowest score (0) represents the absence of pain, while the highest score (10) corresponds to the maximum pain possible.
  Only the final results of the study are reported.
Time Frame: 6 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Rehabilitation | Low Lever Laser Acupuncture
Number analyzed (Participants) | 13 | 13
units on a scale | 2.7 (1.9) | 1.2 (1.4)

ADVERSE EVENTS:
Time Frame: 6 weeks
Arm/Group | Rehabilitation | Low Lever Laser Acupuncture
All-Cause Mortality (participants affected / at risk) | 0/13 | 0/13
Serious Adverse Events (participants affected / at risk) | 0/13 | 0/13
Other Adverse Events (participants affected / at risk) | 0/13 | 0/13

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No